CLINICAL TRIAL: NCT06507176
Title: Comparison of the Efficacy of Flexible Ureteroscope and Percutaneous Nephroscopic Surgery in the Treatment of 2-4cm Kidney Stones: a Multicenter Prospective Randomized Controlled Trial
Brief Title: Comparison of the Efficacy of Flexible Ureteroscope and Percutaneous Nephroscopic Surgery in the Treatment of 2-4cm Kidney Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yanbo Wang, Clinical Professor, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: yanbo wang
Record Dates: First submitted 2024-07-04; First posted 2024-07-18 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Kidney Stone
Keywords: kidney stone; flexible ureteroscope; percutaneous nephroscopic surgery
MeSH Terms: conditions — Kidney Calculi | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flexible ureteroscopic lithotripsy (Experimental)
  Interventions: Procedure: flexible ureteroscopic lithotripsy
- percutaneous nephrolithotomy (Active Comparator)
  Interventions: Procedure: percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: flexible ureteroscopic lithotripsy — This group of patients underwent flexible ureteroscopic lithotripsy.
  Arms: flexible ureteroscopic lithotripsy
Procedure: percutaneous nephrolithotomy — This group of patients underwent percutaneous nephrolithotomy.
  Arms: percutaneous nephrolithotomy

SUMMARY:
Urolithiasis is a common disease in urology. With the continuous progress of science and technology, the treatment of kidney lithiasis has undergone revolutionary changes, and the previously commonly used open surgical lithotomy method has been gradually eliminated, and replaced with less traumatic treatment methods. Percutaneous nephroscopy can theoretically treat the vast majority of kidney stones, especially in the treatment of kidney stones > 2 cm, it is widely used. With the development of ureteroscopy technology, the adaptation of ureteroscopy for the treatment of kidney stones has been expanding, and people have gradually paid attention to it with less damage and higher safety. This study aims to evaluate whether the efficacy and safety of soft ureteral lithotomy in the treatment of 2-4cm kidney stones is equal to that of percutaneous nephrolithotomy through prospective randomized controlled clinical trials, so as to provide more choices for physicians and patients, and provide theoretical basis for the standardization of clinical practice and the rationality of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient agrees to participate in the experiment and signs the informed consent, including compliance with the requirements of the experiment
2. American Society of Anesthesiologists (ASA) score of 1-2, tolerate surgery
3. Age 18-70 years old
4. Diagnosed with renal stones via CT scan, with the largest diameter of the stone being 2-4 cm.

Exclusion Criteria:

1. Excessive obesity, BMI > 28
2. Severe urinary tract infection not corrected
3. Previous history of kidney transplantation or urinary tract diversion surgery
4. Uncorrected bleeding or patients with coagulation dysfunction
5. Urinary system congenital malformations, such as polycystic kidney, horseshoe kidney, pelvic ectopic kidney, etc
6. Combined with serious heart and lung dysfunction and failure of important organs and cannot tolerate anesthesia or surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-07-21 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Stone free-rate (SFR) | All patients underwent a 2mm plain CT scan 1 month after surgery to assess final SFR.
  Stone-free status is defined as the absence of any residual stone fragments or the presence of clinically meaningless residual stone fragments in the kidney, defined as ≤4mm, asymptomatic, non-obstructive, and non-infectious stone particles.

SECONDARY OUTCOMES:
Time of operation | From transurethral surgery to indwelling fistula or catheter, assessed up to 6 hours.
  Time of operation：From transurethral surgery to indwelling fistula or catheter.
Length of stay | From leaving the operating room to discharge,assessed up to 1 month.
  Length of stay: from leaving the operating room to discharge
Postoperative complication | Any surgery-related adverse events that occurred during or less than one month after surgery.
  Postoperative complication：Any surgery-related adverse events that occurred during or less than one month after surgery
Hospitalization costs | From admission to discharge,assessed up to 1 month.
  Hospitalization costs: Total costs during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Yanbowang, Ch’ang-ch’un, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication